CLINICAL TRIAL: NCT05550922
Title: The Effect of Health Care Transition Based Education Program Given to Asthmatic Adolescents on Transition Readiness and Self-Efficacy
Brief Title: The Effect of Health Care Transition Based Education Given to Adolescents With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10742606484
Record Dates: First submitted 2022-09-10; First posted 2022-09-22 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Asthma in Children
Keywords: Adolescents; Transfer to adult care; Transitional care; Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthcare transition based education (Experimental): The content of the education program and interviews include: the importance of transition readiness from pediatric to adult care; asthma, asthma management, asthma support groups and literature; asthma self-management skills (making appointments, taking medications regularly, knowing the risks and what to do during an asthma attack, visiting doctors alone, getting a prescription, communicating with health care professionals); filling out medical forms; insurance; decision making, autonomy, career plans; characteristics of adolescence; pediatrics and adult care differences; transition planning; discussions on case studies; knowledge and skills related to adult pulmonology service procedures; interview with pediatric and adult pulmonologists.
  Interventions: Behavioral: Healthcare Transition-Based Education
- No Intervention (No Intervention): Control: Not all control group participants will receive health care transition-based training. The control group will receive standard outpatient clinic asthma treatment during this process.

INTERVENTIONS:
Behavioral: Healthcare Transition-Based Education — The goal is for asthmatic adolescents to take responsibility for their own disease, be prepared for transition to adult pulmonology services, increase their self-efficacy, and gain management skills as a result of health care transition education.
  Arms: Healthcare transition based education

SUMMARY:
Aim: The purpose of this study was to examine the effect of health care transition-based education on transition readiness and self-efficacy in adolescents (14-18 years) with asthma through a randomized controlled experimental study that integrated the literature, model, and research on the transition from pediatrics to adult care.

The research hypotheses are as follows:

H0: There is no significant difference between the intervention and control groups' mean "Transition Readiness Assessment Questionnaire", "Self Efficacy Scale for Children and Adolescents with Asthma" and "Mind the Gap Scale" scores before and after the education they received on health care transition.

H1: The mean "Transition Readiness Assessment Questionnaire", "Self Efficacy Scale for Children and Adolescents with Asthma" and "Mind the Gap Scale" score of the treatment group is significantly higher than the control group after the education they received on health care transition.

DETAILED DESCRIPTION:
Asthma is one of the most prevalent chronic inflammatory diseases in children, negatively impacting more than 7.5% of those under the age of 18. Data indicate that more than half of children with asthma have asthma management failures, resulting in increased healthcare use. Because childhood asthma is a risk factor for the development of chronic obstructive pulmonary disease later in life, it is critical to keep adolescents on track even if their asthma is mild. Furthermore, despite adolescent remission, asthma can resurface in adulthood. As a result, it is critical to identify the factors influencing the transition from pediatric to adult services and to plan for an appropriate transition. Adolescents are expected to be capable of self-management in their own lives and to be willing to accept responsibility for their own health. However, the disparities in care and approach difference between pediatric and adult services increase adolescent resistance to adult care. Following the transition, many difficulties can arise, including changing the adult doctor, failing to attend regular check-ups, discontinuing medication, increasing the use of emergency rooms, and increasing the cost of care. Furthermore, parents become concerned that their children will be unable to care for themselves during the transition to adult service. Health care transition is the deliberate and planned transfer of chronically diagnosed adolescents and young adults' physical and medical conditions from pediatrics-centered care to the adult health care system. Comprehensive planning and information are essential for reducing their anxiety and uncertainty about the transition. The purpose of this study was to examine the effect of health care transition-based education on transition readiness and self-efficacy in adolescents (14-18 years) with asthma through a randomized controlled experimental study that integrated the literature, model, and research on the transition from pediatrics to adult care. The number of children in the groups will be analyzed based on another study in which one of the scales to be used in the study. According to the calculations made in the G-Power 3.1 Demo package program, when the effect size is accepted as 0.75, it was seen that at least 23 cases in each group would be sufficient for 90% power. Because of the possibility of data loss among the participants, it was planned to recruit a total of 60 adolescents. Following the study, power analysis was carried out using the GPOWER 3.1.7 statistical analysis software. The intervention group: Adolescents with asthma will receive one-on-one training on transitioning from the pediatric to adult care, as well as on asthma self-management skills. After retrieving the written consent from the parents and the adolescents, the trainings will be held every two weeks for a total of six sessions over Zoom for three months. Following each training session, four face-to-face individual interviews will be held in a hospital quiet room. Individual interviews at the hospital have been scheduled to last 30 to 40 minutes, with one-on-one training sessions lasting an average of 40 minutes. The adolescent and parent will receive reminder messages the day before the training sessions and the face-to-face meeting. Not all control group participants will receive health care transition-based training. The control group will receive standard outpatient clinic asthma treatment during this process. Following the completion of the study, a training booklet will be distributed to the children in the control group in a way that does not affect the study data.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 14-18
* Adolescent and parent's consent to participate in the research
* Completing all trainings and follow-ups during the research period.
* Understanding and speaking Turkish
* Having had an asthma diagnosis for at least a year
* Having no mental deficiency that may prevent communication
* Access to internet and a computer

Exclusion Criteria:

* Not being between the ages of 14-18
* Another chronic disease
* Not completing all trainings and follow-ups during the research period.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
The Transition Readiness Assessment Questionnaire (TRAQ) | TRAQ score will evaluate at baseline
  The Transition Readiness Assessment Questionnaire contains a series of questions in which the youth is asked to describe their ability level in various skill areas related to their health and health care, using the following scale: No, I do not know how No, but I want to learn No, but I am learning to do this Yes, I have started doing this Yes, I always do this when I need to. The 1 to 5 likert type scale consists of 20 questions. This produces a minimum score 20, max score 100. A higher score indicates a better outcome.
The Transition Readiness Assessment Questionnaire (TRAQ) | TRAQ score will evaluate at third month
  The Transition Readiness Assessment Questionnaire contains a series of questions in which the youth is asked to describe their ability level in various skill areas related to their health and health care, using the following scale: No, I do not know how No, but I want to learn No, but I am learning to do this Yes, I have started doing this Yes, I always do this when I need to. The 1 to 5 likert type scale consists of 20 questions. This produces a minimum score 20, max score 100. A higher score indicates a better outcome.

SECONDARY OUTCOMES:
Self Efficacy Scale for Children and Adolescents with Asthma (SESCAA) | SESCAA score will evaluate at baseline.
  This scale is divided into three sub-dimensions: asthma-related medical knowledge, asthma management skills, and problem-solving skills. This scale was developed to assess how adolescents and children with asthma make decisions and manage their condition. The 1 to 5 likert type scale consists of 22 questions. Score is 22-110, a higher score indicates a better outcome.
Self Efficacy Scale for Children and Adolescents with Asthma (SESCAA) | SESCAA score will evaluate at third month
  This scale is divided into three sub-dimensions: asthma-related medical knowledge, asthma management skills, and problem-solving skills. This scale was developed to assess how adolescents and children with asthma make decisions and manage their condition. The 1 to 5 likert type scale consists of 22 questions. Score is 22-110, a higher score indicates a better outcome.
Mind the Gap Scale (MGS) | MGS score will evaluate at baseline
  Mind the Gap Scale enables adolescents with chronic diseases to self-evaluate the care they receive and set their own expectations; considers the care provided in terms of "physical environment management", "health personnel characteristics" and "care process"; It is a short scale that is simple to use. It is based on the theory of contradiction, which explains the gap between one's ideals, expectations, and what they actually perceive. Based on this, the difference between the adolescent's expectation of "ideal care" and his or her opinions about current care reflects the patient's level of satisfaction. If the adolescents' views on current care are lower than the "ideal care" scores, they are dissatisfied with the care they are receiving. The 1 to 7 Likert type scale consists of 21 questions. The level of satisfaction decreases as the difference in scores obtained from the scale increases.
Mind the Gap Scale (MGS) | MGS score will evaluate at third month
  Mind the Gap Scale enables adolescents with chronic diseases to self-evaluate the care they receive and set their own expectations; considers the care provided in terms of "physical environment management", "health personnel characteristics" and "care process"; It is a short scale that is simple to use. It is based on the theory of contradiction, which explains the gap between one's ideals, expectations, and what they actually perceive. Based on this, the difference between the adolescent's expectation of "ideal care" and his or her opinions about current care reflects the patient's level of satisfaction. If the adolescents' views on current care are lower than the "ideal care" scores, they are dissatisfied with the care they are receiving. The 1 to 7 Likert type scale consists of 21 questions. The level of satisfaction decreases as the difference in scores obtained from the scale increases.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma DİNÇ, PhD Student, Principal Investigator — Saglik Bilimleri University
Locations (1):
- Gulhane Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dinc F, Yildiz D, Ercan N. The effectiveness of an education program based on healthcare transition in adolescents with asthma: A randomized controlled trial. Pediatr Allergy Immunol. 2024 Mar;35(3):e14101. doi: 10.1111/pai.14101. PMID 38456636